CLINICAL TRIAL: NCT03806816
Title: Use of Melatonin for Neuroprotection in Term Infants With Hypoxic-ischaemic Encephalopathy
Brief Title: Use of Melatonin for Neuroprotection in Asphyxiated Newborns
Acronym: MELPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Collaborators: AUSL Romagna Rimini (Other)
Responsible Party: Principal Investigator, Anna Tarocco, Medical Doctor, Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23/2018/SPER/AOUFE
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Cell Damage; Asphyxia Perinatal
Keywords: autophagy; neuroprotection; melatonin; Hypoxic-Ischemic Encephalopathy; hypothermia; newborn; neurological outcome; perinatal asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYPOTHERMIA / MELATONIN group (Experimental): HIE infants who will receive melatonin in addition to the routine cooling treatment
  Interventions: Dietary Supplement: Melatonin
- HYPOTHERMIA / PLACEBO group (Experimental): HIE infants who will not receive melatonin in addition to the routine cooling treatment
  Interventions: Other: PLACEBO group

INTERVENTIONS:
Dietary Supplement: Melatonin — 5 daily enteral doses of melatonin 10 mg/kg. (=2 ml/kg)
  Other Names: Buona Circadiem
  Arms: HYPOTHERMIA / MELATONIN group
Other: PLACEBO group — 5 daily enteral doses of placebo 2 ml/kg
  Other Names: placebo
  Arms: HYPOTHERMIA / PLACEBO group

SUMMARY:
Protection of brain development is a major aim in the Neonatal Intensive Care Unit. Hypoxic-Ischemic Encephalopathy (HIE) occurs in 3-5 per 1000 births. Only 47% of neonates have normal outcomes. The neurodevelopmental consequences of brain injury for asphyxiated term infants include cerebral palsy, severe intellectual disabilities and also a number of minor behavioural and cognitive deficits. However, there are very few therapeutic strategies for the prevention or treatment of brain damage. The gold standard is hypothermic treatment but, according to the literature, melatonin potentially acts in synergy with hypothermia for neuroprotection and to improve neurologic outcomes. Melatonin appears to be a good candidate because of its different protective effects including reactive oxygen species scavenging, excitotoxic cascade blockade, modulation of neuroinflammatory pathways.

The research study will evaluate the neuroprotective properties and the effects of Melatonin in association with therapeutic hypothermia for hypoxic ischemic encephalopathy.

DETAILED DESCRIPTION:
It is a randomized double blind, placebo controlled trial on 100 neonates with moderate to moderately to severe hypoxic ischemic encephalopathy (HIE) . HIE infants are randomized into two groups: Whole body cooling group (N = 50 receive 72 hours of whole body hypothermia) and melatonin/ hypothermia group (N = 50; receive hypothermia and 5 daily enteral doses of melatonin 10 mg/kg). Serum melatonin and autophagy levels are measured at enrollment, daily during the hypothermic treatment, at day 5 and 7 for the two HIE groups.

aEEG will be performed for 72 hrs during the hypothermic treatment and the re-warming. MRI and Spectroscopy analysis will be performed between day 5 and 7 of. After hospital discharge the infants will enter a follow-up program consisting in periodic clinical and developmental assessments until 2 years of age corrected for prematurity. An expert psychologist and a neonatologist will assess neurodevelopmental outcome using the Bayley Scales III at 6-12-24 months of corrected age.

ELIGIBILITY:
Inclusion Criteria:

* gestational age > 35 weeks and weight > 1800 gr
* Apgar score < 5 at 10 minutes o need for cardiopulmonary resuscitation at 10 minutes or evidence of base excess > 12 mmol/L or pH < 7,0 at initial blood gas analyses
* evidence of moderate or severa encephalopathy graded according to Sarnat&Sarnat neurological evaluation
* abnormal amplitude integrated electroencephalography

Exclusion Criteria:

* suspected inborn errors of metabolism
* major chromosomal congenital defects

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Bayley III scale | 12 months
  Bayley scale of infant and toddler development. It measures developmental skills reached by infant and young children between 1 month and 42 months The scale is subdivided into 5 subscales Cognitive,Receptive communication,Expressive communication,Fine motor ,Gross motor.Receptive and expressive communication have a composite in language score So as fine and gross motor in motor score For all subtests raw scores correspond to scaled scores ranging from 1 to 19 with a mean of 10 and SD of 3 The composite scores are given by the sum of the corresponding subtests scaled scores.
  Two parent-reported scales (Social-Emotional and Adaptive Behavior) will be collected.

SECONDARY OUTCOMES:
brain MRI | between the 5th and 7th days of life
  to evaluate the presence of deep grey matter, PLIC, white matter, brainstem and hippocampus lesions
continuous aEEG | Continuous monitoring for the first 72 hours and for the rewarmed
  Al Naqueeb classification for aEEG will be used.Background voltage pattern will be scored in NORMAL (Lower margin >5μV,Upper margin >10μV The activity is continuous), MODERATELY ABORMAL (Lower margin <5μV, upper margin >10μV,The activity is moderately discontinuous)SEVERELY ABNORMAL/ SUPPRESSED (Lower margin <5μV, upper margin <10μV)
Plasma Concentration of Melatonin | at birth, 24 hours, 48 hours, 72 hours, 5 days, 7 days of life
  UPLC-Massa Acquity-Xevo TQD (Waters) will be used to measure melatonin concentrations in the plasma
ATG5 Plasma concentration | at birth, 24 hours, 48 hours, 72 hours, 5 days, 7 days of life
  ELISA test will be used to measure plasma levels of ATG5

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tarocco, MD, Principal Investigator — University Hospital of Ferrara
Locations (6):
- Ospedale Pediatrico Bambin Gesù, Vatican City, Holy See
- Italy (5):
  - ospdale di Bolzano, Bolzano
  - Bufalini Hospital Cesena, Cesena
  - University Hospital "Sant'Anna" of Ferrara, Ferrara
  - ospedale San Salvatore, L’Aquila
  - Infermi Hospital Rimini, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang Q, Lv H, Lu L, Ren P, Li L. Neonatal hypoxic-ischemic encephalopathy: emerging therapeutic strategies based on pathophysiologic phases of the injury. J Matern Fetal Neonatal Med. 2019 Nov;32(21):3685-3692. doi: 10.1080/14767058.2018.1468881. Epub 2018 May 2. PMID 29681183
- [Result] Hassell KJ, Ezzati M, Alonso-Alconada D, Hausenloy DJ, Robertson NJ. New horizons for newborn brain protection: enhancing endogenous neuroprotection. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F541-52. doi: 10.1136/archdischild-2014-306284. Epub 2015 Jun 10. PMID 26063194
- [Result] McAdams RM, Juul SE. Neonatal Encephalopathy: Update on Therapeutic Hypothermia and Other Novel Therapeutics. Clin Perinatol. 2016 Sep;43(3):485-500. doi: 10.1016/j.clp.2016.04.007. Epub 2016 Jun 22. PMID 27524449
- [Result] Ramos E, Patino P, Reiter RJ, Gil-Martin E, Marco-Contelles J, Parada E, de Los Rios C, Romero A, Egea J. Ischemic brain injury: New insights on the protective role of melatonin. Free Radic Biol Med. 2017 Mar;104:32-53. doi: 10.1016/j.freeradbiomed.2017.01.005. Epub 2017 Jan 6. PMID 28065781
- [Result] Balduini W, Carloni S, Perrone S, Bertrando S, Tataranno ML, Negro S, Proietti F, Longini M, Buonocore G. The use of melatonin in hypoxic-ischemic brain damage: an experimental study. J Matern Fetal Neonatal Med. 2012 Apr;25 Suppl 1:119-24. doi: 10.3109/14767058.2012.663232. Epub 2012 Mar 5. PMID 22348528
- [Result] Parikh P, Juul SE. Neuroprotective Strategies in Neonatal Brain Injury. J Pediatr. 2018 Jan;192:22-32. doi: 10.1016/j.jpeds.2017.08.031. Epub 2017 Oct 12. No abstract available. PMID 29031859
- [Result] Martinello K, Hart AR, Yap S, Mitra S, Robertson NJ. Management and investigation of neonatal encephalopathy: 2017 update. Arch Dis Child Fetal Neonatal Ed. 2017 Jul;102(4):F346-F358. doi: 10.1136/archdischild-2015-309639. Epub 2017 Apr 6. PMID 28389438
- [Result] Shea KL, Palanisamy A. What can you do to protect the newborn brain? Curr Opin Anaesthesiol. 2015 Jun;28(3):261-6. doi: 10.1097/ACO.0000000000000184. PMID 25827279
- [Result] Alonso-Alconada D, Alvarez A, Arteaga O, Martinez-Ibarguen A, Hilario E. Neuroprotective effect of melatonin: a novel therapy against perinatal hypoxia-ischemia. Int J Mol Sci. 2013 Apr 29;14(5):9379-95. doi: 10.3390/ijms14059379. PMID 23629670
- [Result] Fan X, van Bel F. Pharmacological neuroprotection after perinatal asphyxia. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:17-9. doi: 10.3109/14767058.2010.505052. PMID 20695757
- [Result] Cilio MR, Ferriero DM. Synergistic neuroprotective therapies with hypothermia. Semin Fetal Neonatal Med. 2010 Oct;15(5):293-8. doi: 10.1016/j.siny.2010.02.002. Epub 2010 Mar 7. PMID 20207600
- [Result] Aly H, Elmahdy H, El-Dib M, Rowisha M, Awny M, El-Gohary T, Elbatch M, Hamisa M, El-Mashad AR. Melatonin use for neuroprotection in perinatal asphyxia: a randomized controlled pilot study. J Perinatol. 2015 Mar;35(3):186-91. doi: 10.1038/jp.2014.186. Epub 2014 Nov 13. PMID 25393080
- [Result] Fulia F, Gitto E, Cuzzocrea S, Reiter RJ, Dugo L, Gitto P, Barberi S, Cordaro S, Barberi I. Increased levels of malondialdehyde and nitrite/nitrate in the blood of asphyxiated newborns: reduction by melatonin. J Pineal Res. 2001 Nov;31(4):343-9. doi: 10.1034/j.1600-079x.2001.310409.x. PMID 11703564
- [Result] Ahmad QM, Chishti AL, Waseem N. Role of melatonin in management of hypoxic ischaemic encephalopathy in newborns: A randomized control trial. J Pak Med Assoc. 2018 Aug;68(8):1233-1237. PMID 30108392
- [Result] Roohbakhsh A, Shamsizadeh A, Hayes AW, Reiter RJ, Karimi G. Melatonin as an endogenous regulator of diseases: The role of autophagy. Pharmacol Res. 2018 Jul;133:265-276. doi: 10.1016/j.phrs.2018.01.022. Epub 2018 Feb 3. PMID 29408249